CLINICAL TRIAL: NCT03068962
Title: Examination of the Distribution of Nitrate Reducing Bacteria in the Human Oral Cavity
Acronym: REBOC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor of Human Nutrition, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 32/16
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: No Dental Disease; Non-smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- beetroot juice (Experimental): Rinse mouth with low nitrate Buxton mineral water followed by holding 10 ml of beetroot juice for 5 min,
  Interventions: Other: beetroot Juice
- low mineral water (Buxton water) (Experimental): Rinse mouth with low nitrate Buxton mineral water followed by holding 10 ml of low nitrate mineral water in the mouth for 5 min or
  Interventions: Other: Buxton water
- antiseptic mouthwash then beetroot juice (Experimental): Rinse with antiseptic mouthwash before holding 10 ml of beetroot juice in the mouth for 5 min
  Interventions: Other: beetroot Juice; Other: antiseptic mouthwash then beetroot juice

INTERVENTIONS:
Other: beetroot Juice — Beetroot Juice
  Arms: antiseptic mouthwash then beetroot juice; beetroot juice
Other: Buxton water — natural mineral water
  Arms: low mineral water (Buxton water)
Other: antiseptic mouthwash then beetroot juice — Chlorhexidine glocunate
  Arms: antiseptic mouthwash then beetroot juice

SUMMARY:
Dietary nitrate have been shown to have health benefits including lowering blood pressure (Hobbs et al, 2012), improving endothelial function and inhibiting platelet aggregation in healthy humans (Lidder & Webb, 2013). The main sources of dietary nitrate in the human diet are vegetables such as beetroot. Nitrates are converted to nitrites then nitric oxide (NO), following their reduction by commensal oral bacteria and those residing in the gastrointestinal tract (Hord, Tang, & Bryan, 2009; Lidder & Webb, 2013). A recent study has shown following elimination of oral bacteria by the use of a chlorhexidine based antiseptic mouthwash, the conversion of nitrate to nitrite is prevented and this is accompanied by a statistically significant increase in blood pressure in normotensive subjects (Kapil et al., 2013). To date, very few studies have investigated the potential role of these oral bacteria in control of blood pressure and if there are any inter and intra-individual differences in bacterial composition.

DETAILED DESCRIPTION:
Volunteers will be provided with an outline of the study and asked to complete a medical and lifestyle questionnaire (in person, email or over the phone). Potentially suitable participants will be identified and asked to attend a screening session during which the study will be explained in more detail before a consent form is signed. Anthropometric measurements will then be taken such as weight, height and blood pressure. Subjects who meet the inclusion criteria will be invited to a further screening session during which time a dentist will check for dental diseases (e.g. current dental cavities or periodontal infection). The oral bacteria samples will be collected in the morning on site at the Department of Food and Nutritional Sciences (Hugh Sinclair Unit of Human Nutrition) on four visit days (including screening visit).On the day before each study visit the volunteers will need to have a low nitrate diet, refrain from strenuous exercise and alcohol, and drink low nitrate mineral water. They will be required to fast overnight and only drink water. In the morning, they will be asked to refrain from brushing their teeth or using mouthwash.

When they arrive in the unit in the fasted state, they will then be randomised to one of three treatments:

* Rinse mouth with low nitrate Buxton mineral water followed by holding 10 ml of beetroot juice (~6 mmol nitrate) for 5 min,
* Rinse mouth with low nitrate Buxton mineral water followed by holding 10 ml of low nitrate mineral water in the mouth for 5 min or
* Rinse with antiseptic mouthwash before holding 10 ml of beetroot juice in the mouth for 5 min.

After 5 mins of holding low nitrate water or beetroot juice in the mouth, they will then spit the whole mouth rinse into a sterile ice-chilled tube.

To evaluate the nitrate reduction in different areas of the oral cavity, the researchers will put filter paper squares which have been soaked in water or beetroot juice in different areas of their mouth (rear, mid and front tongue, tooth surface, buccal surface, hard palate, and sublingual). Volunteers will be required to keep the filter papers in their mouth for 90 seconds before they are removed.

Finally, the oral bacteria will be collected from the 7 sites by sliding a piece of sterile oral floss between the 2 back molars and by swabbing a micro brush along the buccal cervical margin of premolars and rear, mid, front tongue. Saliva will be obtained using a sterile cotton swab. All samples will be placed into sterile tubes (Eppendorfs). Mouth rinse will be collected in sterile ice-chilled Falcon tubes.

Volunteers will then be provided with a light breakfast before they leave the unit. Facilities will be available for participants to brush their teeth before they leave the clinical unit.

The study visits will be separated by at least 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* A signed consent form
* Age 18-55 years
* Non-smoking, healthy individuals
* BMI 18.5 - 30 kg/m2

Exclusion Criteria:

* Diagnosed with a chronic illness
* Individuals with food allergies or allergies to medicated mouthwash or ingredients in the oral products
* Requirements to take long-term medication active on the oral cavity or taken antibiotics within the last 3 months
* Current diagnosis of dental caries, gingivitis, or periodontal disease or chronic oral complaints or Existing oral pathology (active caries lesions and/or periodontal disease; mucosal lesions; poor occlusion)
* Current smoker (regular and electronic cigarettes and cigars)
* Participating in a dietary intervention study.
* Excessive alcohol consumption (> 21 units/wk male, >14 units/wk female)
* Females who are pregnant or lactating
* Reduced salivary flow (unstimulated flow less than 0.1 ml/min);
* less than four natural (enamel) buccal surfaces of upper molars available;
* presence of fixed or removable oral appliances (e.g., dentures, orthodontic wires)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 10 men and 10 women
Enrollment: 20 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2017-09 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
oral bacteria sample will be collected to Identification of nitrate reductase-positive bacteria in the oral cavity and capacity to reduce dietary nitrate | 1 year
  In vitro method will be used to isolate the nitrate reducing bacteria then 16SrDNA sequencing will be used to identify the species of these bacteria.

SECONDARY OUTCOMES:
Identify the major sites in the human oral cavity which contain nitrate reducing bacteria. | 1 year
  filter paper will be put in different sites around the oral cavity in human trial and then removed before analysis using chemiluminescence to determine nitrate and nitrite concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc, PhD, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Background] Hobbs DA, Kaffa N, George TW, Methven L, Lovegrove JA. Blood pressure-lowering effects of beetroot juice and novel beetroot-enriched bread products in normotensive male subjects. Br J Nutr. 2012 Dec 14;108(11):2066-74. doi: 10.1017/S0007114512000190. Epub 2012 Mar 14. PMID 22414688
- [Background] Hord NG, Tang Y, Bryan NS. Food sources of nitrates and nitrites: the physiologic context for potential health benefits. Am J Clin Nutr. 2009 Jul;90(1):1-10. doi: 10.3945/ajcn.2008.27131. Epub 2009 May 13. PMID 19439460
- [Background] Kapil V, Haydar SM, Pearl V, Lundberg JO, Weitzberg E, Ahluwalia A. Physiological role for nitrate-reducing oral bacteria in blood pressure control. Free Radic Biol Med. 2013 Feb;55:93-100. doi: 10.1016/j.freeradbiomed.2012.11.013. Epub 2012 Nov 23. PMID 23183324
- [Background] Lidder S, Webb AJ. Vascular effects of dietary nitrate (as found in green leafy vegetables and beetroot) via the nitrate-nitrite-nitric oxide pathway. Br J Clin Pharmacol. 2013 Mar;75(3):677-96. doi: 10.1111/j.1365-2125.2012.04420.x. PMID 22882425